CLINICAL TRIAL: NCT01501981
Title: Impact of Therapy Optimization on the Level of Biomarkers in Patients With Acute Decompensated and Decompensated Chronic Heart Failure
Brief Title: Impact of Therapy Optimization on the Level of Biomarkers in Patients With Decompensated Heart Failure
Acronym: MOLITOR
Status: Completed | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Brahms AG (Industry)
Responsible Party: Principal Investigator, Verena Tscholl, Dr. med. univ., Charite University, Berlin, Germany
Other Study IDs: 20120211
Record Dates: First submitted 2011-03-30; First posted 2011-12-30 (Estimated); Last update posted 2017-07-25 (Actual); Status verified 2017-07

CONDITIONS: Decompensated Heart Failure
Keywords: heart failure; MR-proANP; MR-proADM; decompensation; Copeptin; CT-proET1; NT-proBNP
MeSH Terms: conditions — Heart Failure; Diabetes Insipidus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
In this pilot, investigator-initiated multi-centre, multinational, observational study the investigators would like to examine the impact of therapy optimization on the level of biomarkers in patients with acute decompensated and decompensated chronic heart failure.

The primary objective is to determine the best time point for measuring biomarker levels during therapy optimization in patients with decompensation to predict clinical outcomes such as mortality, hospitalisation, and quality of life.

Secondary objectives are:

1. To evaluate the impact of guideline-recommended medication on biomarker levels during and following recompensation.
2. To evaluate whether the trajectory of relevant biomarkers (MR-proANP, MR-proADM) is of relevance to guide medical therapy following decompensation.
3. To evaluate whether the degree of biomarker change (e.g. slow versus rapid change) is of relevance with regard to hemodynamic stability and cardiovascular events such as hospitalisation.
4. To evaluate whether the trajectory of relevant biomarkers (copeptin, CT-pro-ET1) is of relevance to guide medical therapy following decompensation.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients ≥ 18 years.
2. Hospitalized for ADHF or decompensated chronic heart failure. Patients who develop ADHF while hospitalized for another reason are not eligible.
3. The underlying primary etiology for decompensation should be cardiac rather than pulmonary disease. For this study, all of the following must be observable at the time of screening:

   * Dyspnea at rest (sitting or supine) or with minimal exertion (such as talking, eating, etc.) - NYHA III/IV;
   * Pulmonary congestion on physical examination or chest x-ray;
4. Able to begin study within 24 hours from presentation to the hospital, including time spent in the emergency department.
5. Be adequately informed of the nature and risks of the study and give written informed consent prior to study start.

Exclusion Criteria:

1. Acute or suspected acute myocardial infarction (AMI) or troponin levels > 3x the upper limit of normal. at the institution's local laboratory.
2. Cardiogenic shock.
3. Temperature > 38°C (oral or equivalent), sepsis or active infection requiring IV antimicrobial treatment.
4. ADHF due to significant arrhythmias (ventricular tachycardia, bradyarrhythmias with ventricular rate < 45 bpm or atrial fibrillation/flutter with ventricular response of > 150 bpm).
5. Current or planned ultrafiltration, hemofiltration, or dialysis.
6. Significant pulmonary disease (history of oral daily steroid dependency, history of CO2 retention or need for intubation for acute exacerbation, or currently receiving IV steroids), or thoracic cage injury which compromises breathing.
7. Any organ transplant recipient or patients currently listed or admitted for transplantation.
8. Acute myocarditis or hypertrophic obstructive, restrictive, or constrictive cardiomyopathy (not including restrictive mitral valve filling patterns).
9. Women who are pregnant or breastfeeding.
10. Malignant disease with a life expectancy of less than two years.
11. Autoimmune disease.
12. Any condition or treatment of a condition which, in the opinion of the investigator, could interfere with the conduct of the study, or which would unacceptably increase the risk of the patient's participation in the study. This may include, but is not limited to, alcoholism, drug dependency or abuse, other severe mental disorders, epilepsy, or any unexplained episodes of syncope.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with acute decompensated and decompensated chronic heart failure
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2011-02; Primary Completion 2013-12 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Time to first event - all cause death - cardiovascular death - all cause hospitalisation - cardiovascular hospitalisation - hospitalization for heart failure | from study start (day 1) during hosptialisation until second year of follow up
  Time to first event
  * all cause death
  * cardiovascular death
  * all cause hospitalisation
  * cardiovascular hospitalisation
  * hospitalization for heart failure

SECONDARY OUTCOMES:
quality of life | from study start (day 1) during hosptialisation until second year of follow up
  The EuroQoL EQ-5D quality of life scale consists of 5 items scaled 1 to 3 reflecting different dimensions of quality of life and a visual analog scale measuring overall self-rated health.
  The Short Form 36 Health Survey. The Hospital Anxiety and Depression Scale (HADS) consists of 14 items measuring symptoms of anxiety and depression in physically ill patients.
  The ENRICHD Social Support Instrument (ESSI) has been developed as a brief tool for measuring perceived social support in the large randomized ENRICHD study.
Six-minute walk test distance | from study start (day 1) during hosptialisation until second year of follow up
  Six-minute walk test distance will be performed at Visit 1-6 a s well as Follow-up after first and second year.
Echocardiographic parameters | from study start (day 1) during hosptialisation until second year of follow up
  Echocardiography (done within the first seven days from the day of entering the study): dimensions of the left ventricle, wall thickness and EF per Simpson (if it is not possible to determine EF per Simpson in particular cases due to very limited sound conditions, then it could be visually assessed by an experienced echocardiographer), diastolic function of the left ventricle per the American Society of Echocardiography (ASE): mitral Doppler, tissue Doppler, pulmonary vein Doppler.

CONTACTS AND LOCATIONS:
Locations (1):
- Charité Campus Virchow Klinikum-Medizinische Klinik mit Schwerpunkt Kardiologie, Berlin, Germany

REFERENCES:
- [Derived] Veskovic J, Cvetkovic M, Tahirovic E, Zdravkovic M, Apostolovic S, Kosevic D, Loncar G, Obradovic D, Matic D, Ignjatovic A, Cvetkovic T, Posch MG, Radenovic S, Ristic AD, Dokic D, Milosevic N, Panic N, Dungen HD. Depression, anxiety, and quality of life as predictors of rehospitalization in patients with chronic heart failure. BMC Cardiovasc Disord. 2023 Oct 27;23(1):525. doi: 10.1186/s12872-023-03500-8. PMID 37891464
- [Derived] Zelenak C, Chavanon ML, Tahirovic E, Trippel TD, Tscholl V, Stroux A, Veskovic J, Apostolovic S, Obradovic D, Zdravkovic M, Loncar G, Stork S, Herrmann-Lingen C, Dungen HD. Early NT-proBNP and MR-proANP associated with QoL 1 year after acutely decompensated heart failure: secondary analysis from the MOLITOR trial. Biomark Med. 2019 Dec;13(17):1493-1507. doi: 10.2217/bmm-2019-0083. Epub 2019 Oct 29. PMID 31659915
- [Derived] Dungen HD, Tscholl V, Obradovic D, Radenovic S, Matic D, Musial Bright L, Tahirovic E, Marx A, Inkrot S, Hashemi D, Veskovic J, Apostolovic S, von Haehling S, Doehner W, Cvetinovic N, Lainscak M, Pieske B, Edelmann F, Trippel T, Loncar G. Prognostic performance of serial in-hospital measurements of copeptin and multiple novel biomarkers among patients with worsening heart failure: results from the MOLITOR study. ESC Heart Fail. 2018 Apr;5(2):288-296. doi: 10.1002/ehf2.12231. Epub 2018 Feb 24. PMID 29476612